CLINICAL TRIAL: NCT01236456
Title: A Phase II Trial of High-dose Cyclophosphamide for Moderate to Severe Refractory Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: High-dose Cyclophosphamide for Moderate to Severe Refractory Chronic Inflammatory Demyelinating Polyneuropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: I am relocating to Johns Hopkins Medical Center
Sponsor: Stony Brook University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65865
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: chronic inflammatory demyelinating polyneuropathy; cyclophosphamide; autoimmune
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide

SUMMARY:
The primary endpoint of this study is to determine what percentage of patients receiving high-dose Cyclophosphamide may experience a halt in the worsening of their disease or experience improvement of their disease and for how long the benefit may last.

DETAILED DESCRIPTION:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a common and under-recognized peripheral neuropathy that is thought to be immune-mediated. Randomized, placebo controlled clinical trials in CIDP demonstrate benefit from treatment with corticosteroids, plasmapheresis, and IV Ig. However, not all patients respond to these therapies. IV cyclophosphamide, cyclosporine, interferons, total lymphoid irradiation, and mycophenolate mofetil have been proposed as appropriate therapies for refractory patients.

Patients with CIDP often respond to immune-modulating treatment. However, the high rate of relapse and treatment-related side effects result in poor long-term outcomes for many patients. CIDP is assumed to be an autoimmune disease, but the pathogenesis is poorly understood. T cell infiltrates are predominantly CD8, suggesting a T cell mediated process. There is not, however, restricted T cell receptor Vbeta utilization seen in sural nerve biopsies. Immunoglobulin and complement deposits noted on the myelin sheaths support an antibody-mediated process. Antibodies to the P0 myelin protein are seen in a minority of patients. High-dose cyclophosphamide is believed to eradicate both B and T lymphocytes. This therapy does not damage hematopoietic stem cells, which allows for rapid white cell recovery without stem cell rescue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CIDP according to the American Academy of Neurology clinical and electrophysiologic criteria
* Age >18 but < 75 years
* Modified Rankin Scale score of >3 after two standard treatment regimens
* Patient must have a left ventricular ejection fraction of >45%
* Serum Creatinine <3mg/dL
* Willingness to participate in a clinical trial

Exclusion Criteria:

* Patients who are preterminal or moribund
* Patients with active malignancies
* Patients with chromosomal abnormalities or peripheral blood counts suggestive of myelodysplastic syndrome
* Patients with active bacterial or fungal infections requiring oral or intravenous antimicrobials are not eligible until resolution of the infection
* Pregnant women and breast-feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-10; Study Completion 2006-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is to evaluate the response rate of CIDP patients as determined by functional score, change in Summated compound motor action potential and strength, after high-dose cyclophosphamide therapy.

SECONDARY OUTCOMES:
The secondary endpoint of this study is to determine remission duration.

REFERENCES:
- [Result] Gladstone DE, Prestrud AA, Brannagan TH 3rd. High-dose cyclophosphamide results in long-term disease remission with restoration of a normal quality of life in patients with severe refractory chronic inflammatory demyelinating polyneuropathy. J Peripher Nerv Syst. 2005 Mar;10(1):11-6. doi: 10.1111/j.1085-9489.2005.10104.x. PMID 15703014
- [Result] Brannagan TH 3rd, Pradhan A, Heiman-Patterson T, Winkelman AC, Styler MJ, Topolsky DL, Crilley PA, Schwartzman RJ, Brodsky I, Gladstone DE. High-dose cyclophosphamide without stem-cell rescue for refractory CIDP. Neurology. 2002 Jun 25;58(12):1856-8. doi: 10.1212/wnl.58.12.1856. PMID 12084892